CLINICAL TRIAL: NCT05531552
Title: The Role of Clinical Pharmacist in Monitoring Drug Therapy in the Cardiovascular and Coronary Care Units in Libya.
Acronym: BSU
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Collaborators: Medical Center Hospital, libya (Unknown); Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa S.H. Alhomri, BCH.PH & pharmaceutical science, Faculty of Pharmacy, Omar Elmokhtar University, Tobruk, Libya., Beni-Suef University
Other Study IDs: Clinical pharmacist role & ICU
Record Dates: First submitted 2022-08-30; First posted 2022-09-08 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-09

CONDITIONS: Coronary Artery Disease
Keywords: clinical pharmacist role, ICU patients, CAD patients,
MeSH Terms: conditions — Coronary Artery Disease | interventions — Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group I (control group): was collect data without any interference (without clinical pharmacy guidelines).
  Subgroup: 10 outpatient, 25 inpatient, 15 patient in CCU.
- Group II (observation group): application of clinical pharmacy guidelines and management CAD. Subgroup: 10 outpatient, 25 inpatient, 15 patient in CCU.
  Interventions: Drug: clinical pharmacy application

INTERVENTIONS:
Drug: clinical pharmacy application — assessment clinical pharmacist in management of CAD and ICU patients.
  Other Names: Follow-up patients and their drugs, to improve health and reduce morbidity and mortality.
  Groups: Group II (observation group)

SUMMARY:
Assessment of role of clinical pharmacist in decreasing morbidity and mortality among coronary artery disease patients.

DETAILED DESCRIPTION:
- Methodology: Follow-up patients from (A to Z) and their risk factors in all phases of disease (CAD) in groups with advised patients to lose weight, decrease smoking, and take medication on time.

Monitoring drugs to CAD by studying its Pharmacodynamic:

Mechanism of action, therapeutic uses [indication], adverse effect and suitable doses, and drug-drug interactions and contraindications

* The study shows the Compare between the patients in (Medical Center Hospital) with and without guidelines of clinical pharmacy. Were managed all by setting a plan with the cardiologist in Libya.

Follow-up was for the one hundred patients in the three groups {Outpatient, Inpatient, and the patients in Cardio Care Unit - CCU}.

* First subgroup, Outpatient: monitored the drugs used in HTN, DM, and Hyperlipidemia (dyslipidemia) to decrease levels of patients who come to the hospital with IHD; therefore, reduce morbidity. Also, it was followed by measurement of BP twice weekly, test for Blood sugar (glucose level) once monthly, and tests the Low-Density Lipoprotein (LDL) at the cardiologist's request.
* Second subgroup, Inpatient: monitored drugs according to international guidelines of clinical pharmacy to decrease the medication errors and management of the drug of stable angina and protected patients from increasing the problem, myocardial infarction, and reduce rates of entry to CCU.
* Third subgroup, Patients in CCU: Practiced the international roles of clinical pharmacy to monitor drug use to unstable Angina and MI, to decrease mortality in Libya.

  * Method of analysis:

Were monitored one hundred patients and divided into:

• Twenty patients from (outpatient) divided to (10pts.-10pts.). (Ten patients) was written the data collected in accordance with the system adopted at the (Medical Center Hospital).

(Ten patients)They are patients who applied the guidelines of clinical pharmacy to them in (Medical Center Hospital) by recommending cardiologists practice the clinical pharmacy guidelines and tailoring doses.

* 50 of inpatients as outpatient (25pts.-25pts.).
* 30 patients in CCU divided into (15pts.-15pts.).

  - The statistical analysis was the comparison between the two groups:
* The first group of patients was undergoing treatment in the (Medical Center Hospital) without applying guidelines. (10 patients-25pts.-15pts.).
* The second group; are a group of patients undergoing treatment in the (Medical Center Hospital) in accordance with guidelines. (10pts.-25pts.-15pts.).

The comparison was in terms of the rate of survival, the speed of symmetry to heal ( i,e. responsiveness to medications), the rate of complications, and death for both groups.

- The purpose of this review is to summarize the role of clinical pharmacy benefits in all aspects of cardiovascular diseases (CVD) in hospitalized patients.

Managed the risk factors (hypertension, diabetes, dyslipidemia) and Ischemic heart disease by monitoring the common drugs in Libya:

* Diuretics: ACEIs and ARBs for hypertension.
* Insulin and Biguanides (Metformin) for diabetes.
* Statins for dyslipidemia.
* Organic nitrates: CCB, BB, Antiplatelets, Anticoagulant, and Fibrinolytics for ischemic heart disease.

And the summary of the aim of the work is the practice of guidelines of clinical pharmacy to manage coronary artery disease to reduce levels of morbidity and mortality in Libya and to prove the need for the presence of clinical pharmacists in Libyan hospitals.

ELIGIBILITY:
Inclusion Criteria:

- The inclusion criteria were all adults ≥40 years of age, with a diagnosis of CAD.

Exclusion Criteria:

* exclusion criteria were patients with various comorbidities such as liver or kidney disease; patients intake alcohol, cardiac surgery and refusal to give informed consent.

Ages: 41 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Follow-up one hundred patients, in two groups, divided each one into three subgroups {10-Outpatient, 25-Inpatient and 15 patients in Cardio Care Unit - CCU}.
  * The first group of patients was undergoing treatment in the (Medical Center Hospital) without applying clinical pharmacy guidelines. (10 patients-25pts.-15pts.).
  * The second group; are a group of patients undergoing treatment in the (Medical Center Hospital) in accordance with clinical pharmacy guidelines. (10pts.-25pts.-15pts.).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Angina pectoris. | 18 months, from Jan 2021 to June 2022.
  Periodically data collected. [ex: the measurements of blood pressure, glucose blood serum, and LDL - (and taken the average during the period)]. The parameters in the research (angina, response to treatment, complication rate, and mortality) - were quantitatively collected, as the results added to the paper contain the number of patients with details of their complications or the cause of death of patients who died).
  The measuring of FBG level (mg/dl), and (LDL-C) mg/dl - was then performed using a fully automated chemistry analysis instrument by Roche company (Cobas Integra 400 plus). And using specific kits for blood glucose levels (System ID 07-6831-6) and using kits for (LDL-C) (System ID 07-6726-3), Troponin (ng\ml) was performed by using (Beckman coulter - Access 2).
  Angina pectoris was more predominant in patients in group (I); vs. in group (II) with a statistically significant difference.
Responsiveness to medications. | 18 months, from Jan 2021 to June 2022.
  Periodically data collected. [ex: the measurements of blood pressure, diabetes, lipid profile, and weight - (and taken the average during the period)]. The parameters in the research (angina, response to treatment, complication rate, and mortality) - were quantitatively collected, as the results added to the paper contain the number of patients with details of their complications or the cause of death of patients who died).
  Follow-up patients, their clinical state and side effects of medications, Following the number of Hospitalization decreased.
  Responsiveness to medications was significantly higher among patients from the group (II); compared with a control group (I)
The incidence of complications. | 18 months, from Jan 2021 to June 2022.
  The complications are noticeable: myocardial infarctions [Troponin was perpetrated by using by (Beckman coulter)(Access 2) ng\ml], cardiac arrhythmias [by ECG], cardiogenic shock [after MI with HF and low BP], HTN crisis {BP measure, DKA [high blood glucose with (+) positive Ketones.
  Data were collected quantitatively, as the results added to the paper contain the number of patients with details of their complications).
The mortality. | 18 months, from Jan 2021 to June 2022.
  The causes of death are cardiogenic shock, ventricular tachycardia, and myocardial infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa S. alhomri, BCH.PH, Principal Investigator — Bachelor of Pharmaceutical Sciences, Faculty of Pharmacy, Omar Elmokhtar University, Tobruk, Libya.; Raghda S. Hussien, Lecturer, Study Director — Clinical Pharmacy Department, Faculty of Pharmacy, Beni-Suef University, Beni- Suef, Egypt.; Eman K. Abdelall, Professor, Study Director — Organic Chemistry Department, Faculty of Pharmacy, Beni-Suef University, Beni- Suef, Egypt.; Ahmed A. Battah, Professor, Study Director — Critical Care Department, Faculty of Medicine, Cairo University, Cairo, Egypt
Locations (1):
- Beni-suef university, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No